CLINICAL TRIAL: NCT04038177
Title: Superset Strength Training for Time-efficiency - A Randomized Controlled Pilot Study
Brief Title: Superset Strength Training for Time-efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-07-VMI
Record Dates: First submitted 2019-07-18; First posted 2019-07-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Sedentary Lifestyle
Keywords: Resistance training; Muscle strength
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superset strength training (Experimental): This is the experimental group that performs strength training with sets and rest intervals programmed in a superset manner
  Interventions: Behavioral: Superset strength training
- Traditional strength training (Active Comparator): This is the comparator group that engages in strength training with sets and rest intervals programmed in accordance with the recommendations from The American College of Sports Medicine
  Interventions: Behavioral: Traditional strength training

INTERVENTIONS:
Behavioral: Superset strength training — Three weeks of familiarization (two times per week) to the exercises leg-press, bench press, lateral pulldown and seated rows, followed by superset strength training two days per week for 12-weeks. Superset 1 are bench-press and seated rows, and superset 2 are leg-press and lateral pulldown. Each superset is performed three times.
  Arms: Superset strength training
Behavioral: Traditional strength training — Three weeks of familiarization (two times per week) to the exercises leg-press, bench press, lateral pulldown and seated rows, followed by strength training two days per week for 12-weeks. Each exercise is performed for three sets with rest intervals between each set.
  Arms: Traditional strength training

SUMMARY:
Physical inactivity is a global challenge and there is an urgent need to find strategies to increases people's activity levels. Strength training is one of the activities that is recommended to engage in regularly by both the American College of Sports Medicine and the World Health Organization. Understanding how strength training can be done effectively without spending much time could potentially increase people's involvement in strength training, as lack of time often is reported as barrier to training. Superset strength training can potentially be a time-efficient way of strength training, as this training method has been found to take half the time of the traditional ways of training.

The aim of the present study is therefore to compare the effects of superset strength training and traditional strength training on muscular strength, body composition and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* living in Trøndelag
* did not perform weekly strength training during the past 6 months.

Exclusion Criteria:

* any known severe somatic condition (e.g., autoimmune and systemic inflammatory diseases, cancer, severe osteoporosis)
* any known severe psychiatric condition
* other contraindications for heavy resistance training (e.g. shoulder pain).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in muscular strength | 3 months
  Change in one repetition maximum strength (weight in kilograms) for all exercises

SECONDARY OUTCOMES:
Change in body weight | 3 months
  Assessed using a body composition analyzer (i.e. InBody)
Change in muscle mass | 3 months
  Assessed using a body composition analyzer (i.e. InBody)
Change in body composition fat mass | 3 months
  Assessed using a body composition analyzer (i.e. InBody)
Change in body composition BMI | 3 months
  Assessed using a body composition analyzer (i.e. InBody)

OTHER OUTCOMES:
Training load | continuously for 3 months
  Assessed by training diaries
Training volume | continuously for 3 months
  Assessed by training diaries
Perceived exhaustion | continuously for 3 months
  Borg Category Ratio Scale (0-10) - information from training diaries
Participant's experiences with the intervention | 3 months
  Semi-structured focus group interviews with questions regarding the experience participant had during the intervention, questions related to the training program, questions related to motivation and fatigue, questions related to time-efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Vegard moe Iversen, PhD, Principal Investigator — Norwegian University of Science and Technology; Øystein Risa, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iversen VM, Eide VB, Unhjem BJ, Fimland MS. Efficacy of Supersets Versus Traditional Sets in Whole-Body Multiple-Joint Resistance Training: A Randomized Controlled Trial. J Strength Cond Res. 2024 Aug 1;38(8):1372-1378. doi: 10.1519/JSC.0000000000004819. PMID 39072654